CLINICAL TRIAL: NCT06815419
Title: In Forcing Spiritual Care: Enhancing Well-Being and Competency in Psychiatric Nurses
Brief Title: Inforcing Spiritual Care: Enhancing Well-Being and Competency in Psychiatric Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Port Said University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Du Rec no 46
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Well-being; Competence

STUDY DESIGN:
Intervention Model Description: The intervention group was trained using a spiritual care education program meanwhile the control group did not receive any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The control group will not receive the spiritual care education program
- Intervention (Experimental): For eight weeks, the intervention group will participate in a spiritual care education program that aimed to improve their ability to provide spiritual care.
  Interventions: Other: spiritual care education program

INTERVENTIONS:
Other: spiritual care education program — The spiritual care education program to improve nurses ability to provide spiritual care. Education includes; Program orientation, an introduction to spiritual care, the concepts of spiritual care, the significance of spiritual care, the theoretical underpinnings of spirituality in mental health, practical strategies for integrating spiritual care in psychiatric nursing, reflective practice, and self-care for enhancing personal spirituality were all covered in the program's weekly two-hour sessions.
  Arms: Intervention

SUMMARY:
This study was done to evaluate the effectiveness of spiritual care education program in enhancing the well-being and competency of psychiatric nurses.

DETAILED DESCRIPTION:
After explaining the aim of the study, an official permission from the aforementioned psychiatric institutions will acquired to carry out the study. In order to prevent conflicts with regular hospital nursing shifts, the study team had arranged the instructional sessions with the head of nurses. Nursing who fulfilled the qualifying requirements and gave their verbal, informed consent was taken by the researchers. Nurses completed the self-administered data collection sheet. The self-administered questionnaire was completed in 15-20 minutes on average. The pre-test questionnaire was first given to both groups prior to the start of the educational session in order to gather data. The post-test was administered using the same pretest questionnaire.

Intervention of spiritual care education/training program For eight weeks, the intervention group participated in a spiritual care education program that aimed to improve their ability to provide spiritual care. Program orientation, an introduction to spiritual care, the concepts of spiritual care, the significance of spiritual care, the theoretical underpinnings of spirituality in mental health, practical strategies for integrating spiritual care in psychiatric nursing, reflective practice, and self-care for enhancing personal spirituality were all covered in the program's weekly two-hour sessions. Throughout the study period, the control group received no intervention and carried on with their regular nursing practice without any further instruction.

The baseline (pre-intervention) questionnaire was given simultaneously to the intervention and control groups in order to gather data at two different times. A questionnaire measuring spiritual well-being and spiritual care competency was filled out by both groups. The filled surveys were gathered by the study team. Both the intervention and control groups received the immediately post-intervention questionnaire simultaneously, right after the educational program concluded.

ELIGIBILITY:
Inclusion Criteria:

The participants of this study were 98 psychiatric nurses working in previously mentioned psychiatric settings and who fulfilled the following inclusion criteria as both male and female, had one year of experience in psychiatric care, willingness to participate in the study and provide informed consent and did not enroll in any ongoing spiritual care-related training.

Exclusion Criteria:

Nurses refused to participate Nurses not on the full duty

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Spiritual Care Competence | 8 weeks
  The scale was used to evaluate spiritual care competencies. The scale was created and validated in English by Van Leeuwen, Tiesinga, Middel, Post, and Jochemsen (2009). It consists of 27 items total, with six subscales. The scale assesses the following six spiritual-care competencies: communication (2 items), professionalization and improving the quality of care (6 items), personal support and counselling of patients (6 items), referral to other professionals (3 items), attitudes towards patients' spirituality (4 items), and assessment and implementation of SC (6 items).
  There are five points ratings on the Likert scale: strongly disagree, disagree, neutral, agree, and strongly agree. Higher scores indicate higher levels of competence; the total score goes from 27 to 135. The subscales demonstrated good homogeneity with average inter-item correlations >0·25 and strong test-retest reliability. Cronbach's α values for the subdimensions of SC assessment and implementation, professiona

SECONDARY OUTCOMES:
Spiritual Well-Being | 8 weeks
  The Spiritual Well-Being Scale (SWBS) used to measure self-perceived spiritual health. The scale was developed by Ellison and Paloutzian in 1982. The 20-item scale was split into two subscales: existential well-being (EWB), which focused on life satisfaction without necessarily being connected to religion, and had 10 items. Religious well-being (RWB), which reflected a sense of fulfilment and connection with God or a higher power and had 10 items.
  The scale is a 6-point Likert scale with 9 negatively worded items to reduce response biases, ranging from Strongly Disagree to Strongly Agree. Higher scores indicate better spiritual well-being; the scale's total scores range from 20 to 120. Three levels have been established for the SWBS scores: low (20 to 40), moderate (41 to 99), and high (100 to 120). High levels of test-retest reliability and internal consistency were demonstrated by the scale. Cronbach's alpha α = 0.87, 0.78, and 0.89 for the RWB, EWB, and SWBS, respectively, indicat

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Port Said, Egypt

IPD SHARING:
Plan to Share IPD: No